CLINICAL TRIAL: NCT02627131
Title: Autologous Bone Marrow Stem Cell Therapy for Autism: An Open Label Uncontrolled Clinical Trial
Brief Title: Autologous Bone Marrow Stem Cell Therapy for Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBG 003
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Autistic Disorder
Keywords: Autism; Stem Cells
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem cell transplantation (Experimental): 2 intrathecal administrations of autologous bone marrow mononuclear cells at baseline and 3 months afterward
  Interventions: Biological: Autologous Bone Marrow Mononuclear Cells

INTERVENTIONS:
Biological: Autologous Bone Marrow Mononuclear Cells — Transplantation of Autologous Bone Marrow Mononuclear Cells

SUMMARY:
The aim of this study was to evaluate the safety and effectiveness of autologous bone marrow mononuclear stem cells in the management of autism.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the safety and effectiveness of autologous bone marrow mononuclear stem cells in the management of autism of 24 patients at Vinmec International Hospital, Hanoi, Vietnam

ELIGIBILITY:
Inclusion Criteria:

- Confirmed diagnosis of autism according to the Diagnostic and Statistical Manual-IV (DSM-IV) diagnostic criteria for autistic disorder

Exclusion Criteria:

* Epilepsy
* Hydrocephalus with ventricular drain
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections
* Severe psychiatric disorders

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Total Score of Childhood Autism Rating Scale (CARS) | 3 months and 6 months after transplantation
  CARS
Number of adverse events | Through study completion, an average of 6 months
  Examples of adverse events to look for: vomiting, increased hyperactivity, fever, bleeding, hematoma, seizures and neurological deficits

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, MD., PhD., Study Chair — Vinmec Healthcare System
Locations (1):
- Vinmec International Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The data without personal identifiers will be published on Dryad.

REFERENCES:
- [Background] Sharma A, Gokulchandran N, Sane H, Nagrajan A, Paranjape A, Kulkarni P, Shetty A, Mishra P, Kali M, Biju H, Badhe P. Autologous bone marrow mononuclear cell therapy for autism: an open label proof of concept study. Stem Cells Int. 2013;2013:623875. doi: 10.1155/2013/623875. Epub 2013 Aug 25. PMID 24062774